CLINICAL TRIAL: NCT04713813
Title: Effectiveness of Hippotherapy Simulator in Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ayk222
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Ankylosing Spondylitis; Exercise
Keywords: Hippotherapy; occupational therapy; horse; Exercise therapy
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized, single-blind, controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: All evaluations for outcomes will perform by the same experienced physiotherapists who will be blind to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group 1(Exercise via mechanical horse-riding simulator) (Active Comparator): Exercise via mechanical horse-riding simulator; Subjects remained in sitting position for 30 minutes on the simulator during these sessions, with extension of the trunk and stabilization of the pelvis. Feet were placed on the footplates as the simulator produced a rhythmic and repetitive movement similar to a walking horse. The simulator can produce several modes of rhythmic and repetitive motions.
  Interventions: Other: Therapeutic exercise program via hippotherapy mechanical stimulator
- Exercise group 2 (Home exercises) (Active Comparator): Home exercises will be consist of a warm-up, stretching, balance, back walking, fingertip walking exercises, the first of which is shown by the physiatrist or physiotherapist to the patients. These patients will be called twice a month to ask whether they have done the exercises, and the patients whose participation rate is below 80% will be excluded from the study by following the exercise schedule when they come to the physician's control monthly.
  Interventions: Other: Therapeutic home exercise program

INTERVENTIONS:
Other: Therapeutic exercise program via hippotherapy mechanical stimulator — Patients were planned to complete hippotherapy exercises sessions 3 times a week for 12 weeks, each lasting 35 minutes per sessions.
  Arms: Exercise group 1(Exercise via mechanical horse-riding simulator)
Other: Therapeutic home exercise program — Patients were planned to complete home exercises sessions 3 times a week for 12 weeks, each lasting 35 minutes per sessions.
  Arms: Exercise group 2 (Home exercises)

SUMMARY:
Recent studies and meta-analysis showed that different exercise plans had greater benefits than no invention group in improving pain, physical function, and disease activity, especially in some studies that involve ankylosing spondylitis patients receiving home-based exercise. Different kinds of exercises are efficacious and should be recommended to AS patients. But, according to our current knowledge, no clear protocols regarding the effectiveness of hippotherapy in AS patients.

This study aims to investigate the effect of the therapeutic horseback riding therapy via a mechanical simulator on disease-specific outcomes and muscle strength of ankylosing spondylitis patients.

DETAILED DESCRIPTION:
Hippotherapy or therapeutic horseback riding therapy is a form of animal-assisted therapy that uses the horse as a modality that aims to improve postural control, balance, and mobility. With hippotherapy, it is aimed to change the center of gravity by using the movements of the horse and to ensure the adaptation of the trunk and pelvis by developing righting and balance reactions against this new position. Current studies suggest that hippotherapy may be a useful complementary treatment approach for improving balance, fatigue, spasticity, walking, and quality of life in different kinds of disabilities. However, horseback riding therapy itself has some limitations as a treatment due to costs, location, and risks. By its nature horse-riding is too dynamic for patients and requires a large outdoor space. It is believed that a hippotherapy simulator is a therapeutic exercise option for the treatment of thoracolumbar segmental instability and hypo-mobility. Besides complications such as fractures caused by falling are greatly reduced using hippotherapy simulators under proper supervision. Hippotherapy with a mechanical stimulator simulates the motion of a horse as part of a continuous therapy package to provide postural or stability training. This exercise develops unified intuitive stimulation plus motor responses. It engages movement hits that are produced by the machine which mimicking the animal walks: this leads to beneficial consequences.

This prospective clinical study aims to investigate the effect of therapeutic horseback riding therapy via a mechanical simulator on disease-specific outcomes and muscle strength of ankylosing spondylitis patients.

This randomized, single-blind, controlled clinical trial will carry out at the University of Usak/ TURKEY.

This randomized, single-blind, controlled clinical trial will carry out at the University of Usak/ TURKEY. The study will include a total of 60 volunteers who had been diagnosed with AS according to the modified New York criteria. The subjects will be patients who are referred to the outpatient physical therapy center of the Physical Medicine and Rehabilitation Department of the Usak University.

Participants will be allocated to the different treatment groups using the block randomization method. All patients in both groups will continue their ongoing medications. But also, both groups will plan to complete exercise sessions 3 times a week for 12 weeks, each lasting 35 minutes per day.

For Group 1 (horse-riding simulator group), patients will perform a horse riding simulation exercise at speeds of 15km/h, 18km/h, 20km/h, 22km/h, 25km/h, each lasting 5 minutes after warm-up for 5 minutes in each session. Then they will rest for five minutes. For safety, a physiotherapist will be accompanied to the exercises for this group.

For Group 2 (home exercise group) patients will perform home exercises. Home exercises will be consist of a warm-up, stretching, balance, back walking, fingertip walking exercises, the first of which is shown by the physiatrist or physiotherapist to the patients. These patients will be called twice a month to ask whether they have done the exercises, and the patients whose participation rate is below 80% will be excluded from the study by following the exercise schedule when they come to the physician's control monthly.

During the study, if, any subject making any changes to the drug treatment will withdraw from the study.

Evaluations will make before and after treatment. All evaluations will perform by the same experienced physiotherapists who will be blind to the study groups.

Primer outcomes of the study; The Bath AS Disease Activity Index (BASDAI) and Bath AS Disease Functional Index (BASFI) will be used for the activity-related disease, function, and baseline measurements of the participants, respectively.

Quadriceps muscle strength will be measured with the microFET®2 Dynamometer. Bath AS Disease Activity Index (BASDAI): This index, which was developed to evaluate disease activity, consists of 6 VAS measurements. These are fatigue, spine, and peripheral joint pain, sensitivity, and morning stiffness measurements.

Bath AS Disease Functional Index (BASFI): BASFI measures the functional capacity of the patient in the previous week. This index consists of 8 questions about daily activities and 2 questions evaluating the patient's ability to cope with daily life. The degree of difficulty felt by the patient in performing specified tasks is marked on a 10 cm visual analog scale. The average of the total score obtained from 10 questions is calculated for use in the analysis.

Quadriceps muscle strength will be measured with the microFET2 Dynamometer. The wireless microFET®2 Digital Handheld Dynamometer muscle tester is an accurate, portable Force Evaluation and Testing device. It is a modern adaptation of the time-tested art of hands-on manual muscle testing. Measurement Range 0-300 lbs force.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis diagnosis according to the modified New York criteria
* Voluntary participation in the study
* Age 18-45 years
* Regular use of disease-modifying anti-rheumatic drugs (methotrexate, sulfasalazine, and anti-tumor necrosis factor (TNF) agents) at a stable dosage for at least six weeks.

Exclusion Criteria:

* Exercising regularly during the previous six months.
* The presence of severe comorbidity that may affect the kidneys, liver, lungs, and heart such as cardiovascular, pulmonary, orthopedic, and neurological problems.
* Problems that may prevent exercise (uncontrollable hypertension, heart attack or history of coronary revascularization, history of syncope or exercise-related arrhythmia, decompensated Type 1 diabetes mellitus, history of hip and/or knee arthroplasty)
* Having undergone any surgery in the previous 6 months
* Any other neuromuscular disease that may affect the muscles' strength.
* Inability to participate in at least 80% of the exercises

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle strength | At the end of the 12th week of exercise schedule
  Quadriceps muscle strength will be measured with the microFET®2 Dynamometer.
Bath Ankylosing Spondylitis Disease Activity Index | At the end of the 12th week of exercise schedule
  The Bath Ankylosing Spondylitis Disease Activity Index consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions asked of the patient pertaining to the five major symptoms of AS: Spinal pain, Fatigue, Arthralgia, Enthesitis, Morning stiffness severity, Morning stiffness duration.
  The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 score. Scores of 4 or greater suggest suboptimal control of disease. Higher values indicate more active disease.
Bath Ankylosing Spondylitis Disease Functional Index | At the end of the 12th week of exercise schedule
  The ten questions that comprise The Bath Ankylosing Spondylitis Functional Index were chosen with input from patients with Ankylosing spondylitis. The first 8 questions evaluate activities related to functional anatomical limitations due to the course of this inflammatory disease. The final 2 questions evaluate the patients' ability to cope with everyday life.
  A visual analogue scale (with 0 being "easy" and 10 "impossible) is used to answer the questions on the test.
  The mean of the ten scales gives the Bath Ankylosing Spondylitis Functional Index score - a value between 0 and 10.
  A higher score indicates a higher degree of functional limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Y KARAHAN, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation Medical Faculty of Usak University /Turkey
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No